CLINICAL TRIAL: NCT04841525
Title: Autism Biomarker Consortium for Clinical Trials (ABC-CT): Follow-up Study
Acronym: ABC-CT
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Boston Children's Hospital (Other); Duke University (Other); University of California, Los Angeles (Other); University of Washington (Other); Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1509016477_b; U01FD006888 (FDA); U19MH108206 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: During Screening Visits, the Autism Diagnostic Observational Schedule (ADOS) will be administered to confirm diagnosis. Criteria for group inclusion is: diagnosis of Autism Spectrum Disorder based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-G), and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
- Typical Development: Typically Developing (TD) participants from each site will be roughly matched by age and sex to the ASD group.

SUMMARY:
This is a multicenter longitudinal follow-up study to the main study of an a registered already (NCT# ). The Follow-up Study (T4) will assess the Main Study cohort for an additional longitudinal time point approximately 2-5 years after the initial study. Children participating in the Follow-up Study will be approximately 8-16 years old.

The aims of the main study is to identify, develop and validate a set of measures that can be used as stratification biomarkers and/or sensitive and reliable objective measures of social impairment in autism spectrum disorders (ASD) that could serve as markers of long term clinical outcome.

DETAILED DESCRIPTION:
All participants who were initially eligible for the main study will be eligible and invited to return regardless of their participation at T2/T3 or current medication/psychiatric status using an intent-to-treat model. The follow-up study will conduct one additional timepoint with participants who enrolled in the main study.

In the Follow-up Study of the Main Study ABC-CT cohort, the investigators will re-administer the biomarker and clinical batteries 2-5 years after original study enrollment. This will allow the investigators to:

1. Assess long-term stability of the markers, extending the analyses of reliability and consistency from the first phase of the consortium.
2. Perform a more robust assessment of sensitivity to change, taking advantage of a longer developmental window in which participants are expected to exhibit greater clinical progression.
3. Evaluate the longitudinal predictive value of the biomarkers by examining the association of their baseline values with later measures of social function.

ELIGIBILITY:
Inclusion Criteria:

For All Subjects:

* Males and Females Age 6 - 11 (<11:5 at timepoint #1 unless all study procedures will be completed before the participant turns 12.0 and prior approval by the Principal Investigator is obtained).
* Written parental consent obtained prior to any study procedures.
* Participant and parent/guardian must be English speaking.

For TD Participants:

• IQ 80-150 as assessed by the Differential Ability Scales (DAS)- 2nd Edition

For ASD Participants:

* Diagnosis of ASD based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5), the Autism Diagnostic Observation Schedule (ADOS-2), and the Autism Diagnostic Interview-Revised, short form (ADI-R). Diagnostic evaluations will be completed by research staff and supervised by a licensed psychologist.
* IQ 60-150 as assessed by the Differential Ability Scales (DAS)- 2nd Edition
* If parents are biological, a minimum of the child and one parent (if accompanying the child at study visits) will be required to participate in the blood draw procedure. It is preferred that the child and both biological parents participate in the blood draw procedure, but the inability to obtain blood samples from trios will not be exclusionary.

Exclusion Criteria:

For All Subjects:

* Known genetic or neurological syndrome with established link to autism (in addition to ASD for ASD participants), but not events in which the link to ASD is less well known/established (e.g., 16p11.2 CNVs, CHD8 mutations, Trisomy 21, 22q deletion syndrome)
* History of epilepsy or seizure disorder (except for history of simple febrile seizures or if the child is seizure free (regardless of seizure type) for the past year).
* Motor or sensory impairment that would interfere with the valid completion of study measures including significant hearing or vision impairment not correctable by a hearing aid or glasses/contact lenses. Children who wear bifocal or progressive lenses are not eligible.
* Medication is not exclusionary. Children taking neurological or psychiatric medications, including anti epileptics and psychopharmacological agents, must be stable on the medication and dose for 8 weeks prior to T1D1.
* History of significant prenatal/perinatal/birth injury (birth <36 weeks AND weight <2000 grams (approximately 4.5lbs)).
* History of neonatal brain damage. (e.g., with diagnoses hypoxic or ischemic event)
* Any other factor that the investigator feels would make assessment or measurement performance invalid.

For ASD Participants:

• Any known environmental circumstances that is likely to account for the picture of autism in the proband (severe nutritional or psychological deprivation etc.)

For TDs Participants:

* Known historical diagnosis of ASD or a sibling with ASD.
* Active psychiatric disorder (depression, anxiety, ADHD, etc.) and/or any current treatment (medication or other treatment) for a psychiatric condition. Participants will be screened using the Child/Adolescent Symptom Inventory (CASI-5). Due to the measurements sensitivity, any score in the clinical range will be reviewed by research staff for determination of eligibility.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 children with an autism spectrum disorder between 6-11 years old, and 75 typically developing children
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
N170 Latency to Upright Human Faces | 5 years
  The N170 Latency to Upright Human Faces (N170 latency) is a scalp recorded EEG event-related potential (ERP) component elicited by perception of the upright human face. Recorded over the posterior-temporal right hemisphere, the latency (or speed) of the peak of the N170 ERP component occurs at approximately 200 msec in children aged 6 to 11 years of age.
Oculomotor Index of Gaze to Human Faces (OMI) | 5 years
  Onscreen gaze position data, reflected in percentage of foveation (angling of the eyes to focus on a particular object) to human faces (Face%) relative to total valid foveation time across three assays.
VABS: Vineland Adaptive Behavior Scales- III Socialization | 5 years
  Administered in person visit during T4D1 or parent phone interview. The Socialization score is based on 3 subdomains of Interpersonal Relationships, Play & Leisure, Coping Scales. The V-Scaled scores, which are specifically designed to measure change over time, are only available for the subdomains. The primary norm-referenced scores for the subdomains are v-scale scores, which have a mean of 15 and standard deviation (SD) of 3. The Vineland-3 is a standardized measure of adaptive behavior--the things that people do to function in their everyday lives.

CONTACTS AND LOCATIONS:
Overall Officials: James McPartland, PhD, Principal Investigator — Yale University Child Study Center
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes